CLINICAL TRIAL: NCT03535766
Title: An Analysis of Treatment Timelines for Lung Cancer Patients Across System Evolutions
Acronym: TRACE
Status: Completed | Type: Observational
Sponsor: St Elizabeth Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: 2/2018-014
Record Dates: First submitted 2018-05-07; First posted 2018-05-24 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a single center, minimal risk, physician initiated retrospective chart review. An analysis of treatment timelines for patients diagnosed with lung cancer within the St. Elizabeth system from January 2013 until study completion. The study investigator and designee(s) will review patient electronic medical records, extracting data related to the symptom presentation, diagnosis, and treatment of new diagnoses of lung cancer. Collected data will focus on dates of encounters, diagnostic imaging/procedures, and treatments, with data analysis evaluating time between care encounters and potential delays in care. The data will be further stratified based on system-wide changes implemented to improve efficiency, patient outcomes, and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen within the St. Elizabeth system
* >=18 years of age
* New diagnosis of histologically or cytologically documented primary lung cancer diagnosed January 2013 or later

Exclusion Criteria:

* Patients with metastatic lung disease of other primary
* Other malignancies at investigator's discretion
* Patient received treatment at a facility outside of St. Elizabeth where records are not available through EPIC
* Patient currently undergoing treatment for new diagnosis of lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with lung cancer within the St. Elizabeth system from January 2013 until study completion.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Time from presentation to treatment | from initial patient presentation with symptoms or incidental finding to first day of treatment, up to 3 years
  Time from initial patient presentation with symptoms or incidental finding to first day of treatment, measured in days.

SECONDARY OUTCOMES:
Additional time between imaging and physician referrals | From identification of concerning nodule to specialist appointment, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Royce Calhoun, MD, Principal Investigator — St Elizabeth Healthcare
Locations (1):
- St. Elizabeth Healthcare, Edgewood, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diaconescu R, Lafond C, Whittom R. Treatment delays in non-small cell lung cancer and their prognostic implications. J Thorac Oncol. 2011 Jul;6(7):1254-9. doi: 10.1097/JTO.0b013e318217b623. PMID 21610526
- [Background] Van de Vosse D, Chowdhury R, Boyce A, Halperin R. Wait Times Experienced by Lung Cancer Patients in the BC Southern Interior to Obtain Oncologic Care: Exploration of the Intervals from First Abnormal Imaging to Oncologic Treatment. Cureus. 2015 Sep 22;7(9):e330. doi: 10.7759/cureus.330. PMID 26543688
- [Background] Vidaver RM, Shershneva MB, Hetzel SJ, Holden TR, Campbell TC. Typical Time to Treatment of Patients With Lung Cancer in a Multisite, US-Based Study. J Oncol Pract. 2016 Jun;12(6):e643-53. doi: 10.1200/JOP.2015.009605. Epub 2016 May 3. PMID 27143146